CLINICAL TRIAL: NCT00046306
Title: Nevada Environmental Tobacco Smoke and Health Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 9520-CP-001
Record Dates: First submitted 2002-09-26; First posted 2002-09-30 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Cardiovascular Disease; Cancer
Keywords: Oxidative Stress; Cardiovascular Disease; Cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms | interventions — Antioxidants

INTERVENTIONS:
Drug: Antioxidants

SUMMARY:
Workplace exposure to secondhand cigarette smoke or environmental tobacco smoke (ETS)is widespread, effecting between 19 and 49% of the U.S. workforce. The first part of this study is designed to test whether exposure to ETS in the workplace effects a person's risk of developing chronic diseases such as cardiovascular disease and cancer. The second part of this study is designed to test whether antioxidant supplementation in this group of ETS exposed individuals can reduce their risk of developing chronic disease.

The study will look at 375 non-smokers who either work on a casino floor or as bartenders or cocktail servers. Initial baseline data will be collected (questionnaires and blood samples taken) and the subjects will be randomized into one of three groups, placebo, low antioxidant supplementation and high antioxidant supplementation. They will be followed over a two-year period, coming in for follow-up testing every six months. Statistical analysis will be conducted to see whether this group of ETS exposed individuals has a greater risk of developing chronic disease and whether the use of antioxidant supplements can moderate any risks.

ELIGIBILITY:
Inclusion Criteria:

Non-smoker Work in a casino - on the casino floor or work as a bartender or cocktail server for at least 1 year Do not take antioxidant supplements Healthy - not diagnosed with any major chronic diseases.

Exclusion Criteria:

Blood pressure SBP>200,<85 DBP>100, <40 Pulse >120, <45 Cholesterol >400 Triglycerides >700 Blood Cotinine >10 ng/ml BMI >35

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375
Dates: Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris A Pritsos, Ph.D., Principal Investigator — University of Nevada, Reno
Locations (1):
- ETS Clinic, University of Nevada, School of Medicine, 1707 W. Charleston Blvd Suite 100, Las Vegas, Nevada, United States